CLINICAL TRIAL: NCT03490409
Title: Effect of Compression Therapy on Postoperative Swelling and Pain, Among Patients With a BMI ≥30 kg/m2, After Total Knee Arthroplasty: A Randomized Controlled Pilot Study
Brief Title: Effect of Compression Therapy on Postoperative Swelling and Pain After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Linda Mie Christensen, Nurse, Naestved Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SJ-635
Record Dates: First submitted 2017-12-01; First posted 2018-04-06 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Edema
Keywords: Arthroplasty; Replacement; Knee; Compression; Edema; Pain
MeSH Terms: conditions — Edema; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- compression stocking (Experimental): The intervention group will receive a thigh compression stocking, which is to be used for 24 hours a day for 14 days after surgery.
  Interventions: Device: Thigh compression stocking
- Conventional treatment (No Intervention): The control group will receive conventional treatment, a compression bandage placed at the end of surgery and removed on the night of the surgery.

INTERVENTIONS:
Device: Thigh compression stocking — Thigh compression stocking
  Arms: compression stocking

SUMMARY:
The number of severely obese patients who has knee replacement surgery is rising. Obesity increases the risk of the postoperative swelling. A complication which can cause pain and discomfort as well as complicate and prolong rehabilitation.

The aim of the present pilot study is to examine the effect of a compression stocking on postoperative swelling and pain among patients with a BMI ≥30 kg/m2, after total knee arthroplasty. The hypothesis is that the use of a medical elastic compression stocking for 14 days postoperatively may reduce postoperative swelling by two cm.

The pilot study will furthermore provide useful information for feasibility which will be used to decide whether or not a larger study should be initiated.

DETAILED DESCRIPTION:
In Denmark approximately 9000 knee replacements were performed in 2015. Almost 7000 of the procedures performed were total knee arthroplasties.

A total knee arthroplasty is a common procedure performed as treatment for knee arthritis.

In 2015, 39,9% of the patients in Denmark who had knee replacement surgery were severely obese with a BMI ≥30 kg/m2.

The percentage of severely obese patients who has knee replacement surgery is rising and studies have shown that obesity increases the risk of postoperative complications.

A danish cross-sectional study found that swelling with a prevalence of 90,7% was the most frequent patient-reported complication after knee arthroplasty. A common postoperative complication after total knee arthroplasty and severe obesity increases the risk of postoperative swelling.

Postoperative swelling may impair movement of the knee, cause pain and discomfort as well as complicate and prolong rehabilitation.

Despite that a BMI 30 kg/m2 causes more postoperative complications, obese patients experience the same quality of life and improvement of function after total knee arthroplasty as patients with a BMI ≤30 kg/m2. The higher complication rate among the obese patients has socioeconomic consequences due to readmission and unscheduled outpatient visits.

A study found that in the first 30 days postoperative after total knee arthroplasty 2,9 percent of the patients were readmitted. In 2015 7,3% of the patients who had primary knee replacement surgery in Denmark were readmitted within 30 days after the operation. Unscheduled outpatient visits 30 days post-surgery, is related to swelling in the operated leg. There is a need for further research on interventions that may prevent postoperative swelling after knee replacement surgery. A compression stocking is a feasible intervention and an effective treatment in the prevention of swelling. The stocking provides measured pressure against the leg which helps the blood to move up toward the heart. By improving the blood flow, swelling is prevented and reduced.

A Danish randomized controlled study (RCT), that investigated the effect of a compression stocking when used for four weeks postoperatively found that the stocking did not have a clinical effect on postoperative swelling.

However the stocking was the day after the surgery, where seventy percent of the postoperative swelling already had occurred.

Therefore it is relevant to investigate whether a compression stocking has an effect on postoperative swelling, when applied immediately after the operation has ended.

The aim of the present pilot study is to examine the effect of a compression stocking on postoperative swelling and pain among patients with a BMI ≥30 kg/m2, after total knee arthroplasty. The aim of the pilot study is furthermore to provide useful information for feasibility which will be used to decide whether or not a larger RCT should be initiated.

All patients will be recruited at Department for planned Orthopaedic Surgery, Naestved Hospital, Denmark.

Inclusion criteria: planned for total knee arthroplasty, BMI ≥30 kg/m2, aged 18 or older, speaks, reads and understands danish and written informed consent.

Collaborating researchers and departments :

Department for Planned Orthopaedic Surgery, Ringstedgade 61, Naestved Hospital, Denmark.

Odense Patient data Explorative Network, J.B. Winsloew Vej 9a, 3. Sal, 5000 Odense C, Denmark

44 patients will be included in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Planned for total knee arthroplasty
* BMI ≥30 kg/m2, aged 18 or older
* Speaks, reads and understands Danish
* Written informed consent.

Exclusion Criteria:

* Peripheral Arterial Disease
* Arterial insufficiency
* No palpable puls at the arteria dorsalis pedis
* Severe atherosclerosis
* Leg ulcers
* Skin disease
* Fragile "tissue paper" skin
* Neuropathy or other cause of sensory impairment
* Allergy to the stocking material
* Massive leg edema or pulmonary edema from congestive cardiac failure,
* Deformity of the leg or unusual leg shape or size preventing correct fit
* Patient that cannot cooperate. For example does not understand the concept of Visual Analogue Scale (VAS) or is not able to use the compression stocking
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Swelling of the knee after operation | Assessment of swelling of the knee from baseline and 1, 2, 14 days after surgery
  Measurements will be taken on the day of admission before surgery and at day 1, 2 and 14 days after surgery in millimeters to determine whether swelling has occurred. No predetermined higher or lower values. Higher values represent a worse outcome. Lower values represents a better outcome.

SECONDARY OUTCOMES:
Swelling of the calf after the operation. | Assessment of swelling of the calf from baseline and 1, 2, 14 days after surgery
  Measurements will be taken on the day of admission before surgery and at day 1, 2 and 14 days after surgery in millimeters to determine whether swelling has occurred. No predetermined higher or lower values. Higher values represent a worse outcome. Lower values represents a better outcome.
Swelling of the ankle after the operation. | Assessment of the swelling of the ankle from baseline and 1, 2, 14 days after surgery
  Measurements will be taken on the day of admission before surgery and at day 1, 2 and 14 days after surgery in millimeters to determine whether swelling has occurred. No predetermined higher or lower values. Higher values represent a worse outcome. Lower values represents a better outcome.
Pain after the operation. | Assessment of pain from baseline and 1, 2, 14 days after surgery
  Measurements will be taken on the day of admission before surgery and at day 1, 2 and 14 days after surgery using Visual Analogue Scale. A pain measurement scale. Minimum score is 0 and maximum score is 100. Higher values represent a worse outcome. Lower values represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mie Christensen, nurse, Principal Investigator — Naestved Sygehus
Locations (1):
- Department for planned Orthopaedic Surgery, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: Undecided